CLINICAL TRIAL: NCT03632213
Title: A Randomized Clinical Trial to Evaluate the Effects of Losartan on Cardiovascular Disease in Patients With Mucopolysaccharidoses IV A and VI
Brief Title: Evaluation of Losartan on Cardiovascular Disease in Patients With Mucopolysaccharidoses IV A and VI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: The Isaac Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-0685
Record Dates: First submitted 2018-08-03; First posted 2018-08-15 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Mucopolysaccharidosis IV A; Mucopolysaccharidosis VI; Mucopolysaccharidoses; MPS IV A; MPS VI; MPS - Mucopolysaccharidosis; Morquio A Syndrome; Morquio Syndrome A; Morquio Syndrome
Keywords: Mucopolysaccharidoses; Losartan; Aortic root dilatation; Echocardiogram; MPS IV; MPS VI
MeSH Terms: conditions — Mucopolysaccharidosis IV; Mucopolysaccharidosis VI; Mucopolysaccharidoses | interventions — Losartan

STUDY DESIGN:
Intervention Model Description: Experimental group: 15 patients, both sexes, will receive Losartan 25 mg orally for 12 months.
  Control group: 15 patients, both sexes, will receive oral placebo for 12 months.
  Eligible research participants for treatment will be randomly assigned to a treatment group or a control group in a ratio of 1: 1. The groups will be stratified by age and type of MPS in the following strata:
  A) Diagnosis of MPS IVA: 20 patients expected B) Diagnosis of MPS VI: 10 patients expected
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan (Active Comparator): Losartan group: 15 patients, both sexes, will receive Losartan 0.4 to 1.4 mg/kg/day orally for 12 months.
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator): Placebo group:15 patients, both sexes, will receive oral placebo for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — Losartan group: 15 patients, both sexes, will receive Losartan 0.4 to 1.4 mg/kg/day orally for 12 months.
  Arms: Losartan
Drug: Placebo — Placebo group: 15 patients, both sexes, will receive oral placebo for 12 months.
  Arms: Placebo

SUMMARY:
Mucopolysaccharidoses (MPS) are multisystemic diseases with significant clinical overlap between their types, with cardiac problems being among the most commonly observed manifestations and are also among the main causes of mortality in these patients. For some of the cardiovascular manifestations, such as aortic root dilation and valve diseases, there is no effective treatment currently available. Losartan, on the other hand, has been shown to be an effective drug for dilation of the aortic root, at least in animal models. This study aims to evaluate the safety and efficacy of losartan in patients with MPS VI and other mucopolysaccharidoses.

DETAILED DESCRIPTION:
Mucopolysaccharidoses (MPS) are a group of lysosomal diseases characterized by deficiency of enzymes responsible for the degradation of glycosaminoglycans. MPS are multisystemic diseases with significant clinical overlap between their types, with cardiac problems being among the most commonly observed manifestations and are also among the main causes of mortality in these patients. Enzyme replacement therapy and bone marrow transplantation, despite being well established treatments, are not yet capable of reversing or preventing the progression of some of the cardiological manifestations of MPS. On the other hand, these patients may benefit from other conventional drug or surgical treatment, which can be instituted at an appropriate time if there is a better understanding of how these manifestations progress. In particular, the occurrence of aortic root dilation, although described in animal models, has only recently been evaluated in the studies on mucopolysaccharidoses.

In addition, verifying the effectiveness of losartan in controlling these manifestations in the animal model opens the perspective of clinical use of this drug. Losartan is a low-cost drug and, if its efficacy is demonstrated, may represent an accessible therapy directed at the unmet needs of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed biochemical or molecular diagnosis of MPS VI or MPS IVA.
* Age between 10 and 40 years.
* Presence of aortic root diameter greater than 1.0 standard deviation, as determined by local measurement.
* Be in a stable treatment regime in the last 3 months (without performing Enzyme replacement therapy (ERT), or performing ERT on a regular basis).
* Patient who agree to participate in the study protocol by signing a free informed consent form.

Exclusion Criteria:

* Patient who underwent previous aortic surgery.
* Patient with aortic root diameter greater than 5 cm.
* Patient on angiotensin-converting-enzyme (ACE) inhibitor. In case of use of beta-blocker, or calcium channel blocker, patient without adequate control of blood pressure in the last 3 months.
* Patients with previous adverse events related to treatment with losartan or contraindication to this treatment.
* Inability, in the opinion of the investigator, to complete the study procedures.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2023-05-04 (Estimated); Study Completion 2023-08-03 (Estimated)

PRIMARY OUTCOMES:
Adverse events related to losartan use | 12 months
  The frequency of adverse events after 12 months will be compared among the groups

SECONDARY OUTCOMES:
Z score of maximal aortic root diameter measured by Valsalva sinus | 12 months
  Reduction over time in the Z score of maximal aortic root diameter measured by Valsalva sinus echocardiogram between the baseline assessment and 12 months after treatment with losartan.
Changes of serum levels of transforming growth factor (TGF-Beta-1) | 12 months
  Changes of serum levels of transforming growth factor (TGF-Beta-1) between baseline and 12 months
Changes of serum levels of brain-type natriuretic peptide (BNP) | 12 months
  Changes of serum levels of brain-type natriuretic peptide between baseline and 12 months
Changes of serum levels of N-terminal pro b-type natriuretic peptide (NT-ProBNP) | 12 months
  Changes of serum levels of N-terminal pro b-type natriuretic (NT-ProBNP) peptide between baseline and 12 months
Changes of serum levels of creatine kinase-myocardial ban (ck-mb) | 12 months
  Changes of serum levels of creatine kinase-myocardial ban (ck-mb) between baseline and 12 months
Changes of serum levels of Chemokine (C-X-C motif) ligand 6 (CXCL6) | 12 months
  Changes of serum levels of Chemokine (C-X-C motif) ligand 6 (CXCL6) between baseline and 12 months
Changes of serum levels of Chemokine (C-X-C motif) ligand 16 (CXCL16) | 12 months
  Changes of serum levels of Chemokine (C-X-C motif) ligand 16 (CXCL16) between baseline and 12 months
Changes of serum levels of Endocan-1 (ESM-1) | 12 months
  Changes of serum levels of Endocan-1 (ESM-1) between baseline and 12 months
Changes of serum levels of Placental growth factor (PLGF) | 12 months
  Changes of serum levels ofPlacental growth factor (PLGF) between baseline and 12 months
Changes of serum levels of Fatty acid binding protein 3 (FAPB3) | 12 months
  Changes of serum levels of Fatty acid binding protein 3 (FAPB3) between baseline and 12 months
Changes of serum levels of Fatty acid binding protein 4 (FAPB4) | 12 months
  Changes of serum levels of Fatty acid binding protein 4 (FAPB4) between baseline and 12 months
Changes of serum levels of Oncostatin M | 12 months
  Changes of serum levels of Oncostatin M between baseline and 12 months
Changes of serum levels of Troponin I | 12 months
  Changes of serum levels of Troponin I between baseline and 12 months
Changes of ventricular-vascular coupling measures as assessed by echocardiography between the baseline and 12 months. | 12 months
  Reduction over time in the ventricular-vascular coupling measures as assessed by echocardiography between the baseline and 12 months.
Changes in mitral valve regurgitation | 12 months
  Alteration of the parameter of mitral valve regurgitation as assessed by a semi-quantitative echocardiographic method between the baseline and 12 months.
Changes in aortic valve regurgitation | 12 months
  Alteration of the parameter of aortic valve regurgitation as assessed by a semi-quantitative echocardiographic method between the baseline and 12 months.
Changes in ejection fraction | 12 months
  Alteration of the ejection fraction measurement as assessed by echocardiography between the baseline and 12 months.
Changes in left ventricular longitudinal strain | 12 months
  Alteration of the measurement of left ventricular longitudinal strain as assessed by echocardiography between the baseline and 12 months.
Changes in E/A ratio | 12 months
  Alteration of the parameter E/A ratio as assessed by echocardiography between the baseline and 12 months .
Changes in E/e' ratio | 12 months
  Alteration of the parameter E/e' ratio as assessed by echocardiography between the baseline and 12 months.

OTHER OUTCOMES:
Glycosaminoglycan after 6 months | 6 months
  Difference in urinary glycosaminoglycan levels after 6 months
Glycosaminoglycan after 12 months | 12 months
  Difference in urinary glycosaminoglycan levels after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Giugliani, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre; Guilherme Baldo, PhD, Study Director — Hospital de Clinicas de Porto Algre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided